CLINICAL TRIAL: NCT02151279
Title: Safety of Chitosan as Wine Fining Agent in Shrimp Allergic Patients
Acronym: SWAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Aveiro University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SWAP study
Record Dates: First submitted 2014-05-20; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Shellfish Allergy
Keywords: Shrimp allergy; Chitosan; fining agent
MeSH Terms: conditions — Shellfish Hypersensitivity | interventions — Chitosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): Chitosan as wine fining agent
  Interventions: Other: Control
- Shrimp allergic patients (Active Comparator): Chitosan as wine fining agent
  Interventions: Other: Chitosan as wine fining agent

INTERVENTIONS:
Other: Chitosan as wine fining agent — The possibility of allergic reactions attributed to traces of chitosan used as a fining agent in wine has not been ruled out, particularly in shrimp allergic patients to whom small traces of the potential allergen may be enough to trigger anaphylactic reactions.
  Arms: Shrimp allergic patients
Other: Control
  Arms: control group

SUMMARY:
Chitosan, the main component of the exoskeletons of crustaceans, mollusks and cephalopods, has been used as a fining agent in wines. However, its safety among patients allergic to shellfish has never been evaluated.

Adult patients followed at the Allergy and Clinical Immunology Department who have been diagnosed with anaphylaxis to shrimp will be invited to participate in the study.

Clinical data will be collected to ascertain for eligibility and written information will be provided. After signing informed consent, included subjects will perform skin prick-to-prick tests (PTP) with shrimp boiling water condensate and with fined and unfined wines. All will perform double blind oral challenge with the fined and unfined wines during 1visit day; the placebo (unfined wine) and active challenge (fined wine with chitosan) will be separated by 2 hours. Challenge protocol will be performed with successive increasing doses administered in 4 steps at 15-minute intervals for a total of 100 mL. During the challenge signs and symptoms will be monitored by a trained physician.

Results will be presented as negative or positive (defined by presence of symptoms and signs of an allergic reaction).

Categorical data will be compared by chi-square test. P<0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Hypersensitivity reactions to wine have been rarely reported in the literature, and they are mainly attributed to grape proteins [1], biogenic amines, salicylates, sulfites or yeast [2,3]. However, wine production traditionally involves fining, during which some ingredients such as tannins are removed by co-precipitation with proteins derived from milk (casein, potassium caseinate), egg (ovalbumin, lysozyme), fish (isinglass) or shrimp (chitosan). These proteins are derived from animal sources which are known to play a role in food allergy. This is an increasingly prevalent health problem in Western countries [4,5] and it may manifest itself as life-threatening anaphylactic shock in the presence of only traces of the allergen. Recently, the safety for wine-fining agents derived from milk, fish and egg was established [6]. However, for chitosan, no studies of its safety as a fining agent in allergic patients were performed until now. Chitosan is used as fining agent by the mead and wine industry because of its electrostatic positive charge. Chitosan is obtained by the deacetylation of Chitin [C8H13NO5N]n , a derivative of glucose, and one of the most common polymers found in nature. It is the main component of the cell walls of some fungi, the exoskeletons of arthropods such as crustaceans and insects, the radulae of mollusks, and the beaks of cephalopods, including squid and octopuses [7].

Seafood plays an important role in human nutrition and health, and Portugal is the European country with the second highest consumption [4]. The prevalence of crustacean allergy seems to vary largely between geographical locations, but it seems common in Portugal [8]. The major shellfish allergen is tropomyosin although other allergens may play an important part in allergenicity. The possibility of allergic reactions attributed to traces of chitosan used as a fining agent in wine has not been ruled out, particularly in shrimp allergic patients to whom small traces of the potential allergen may be enough to trigger anaphylactic reactions. Our aim is, therefore, to establish the safety of wine containing chitosan in patients who are severely allergic to shrimp [9].

Potential Risks Several studies published in the literature have evaluated the safety of skin tests, but mostly using commercial extracts. Prick-tests to native foods, called prick-to-prick tests, have been less extensively studied. The CICBAA1 data, from 1,138 food allergic patients of all ages, cover 34,905 prick-to-prick tests to foods. The risk of systemic reactions was evaluated at 0.008% [10, 11]. The negative predictive accuracy for skin prick testing to foods is uniformly high. A negative skin test confirms the absence of an IgE-mediated reaction with 90 to 95% accuracy [12,13]. Therefore, skin testing is highly useful for excluding IgE-mediated food allergy.

However, when positive, these tests, which evaluate sensitization and not clinical allergy, are not without pitfalls, and their results must be confirmed by an oral challenge to avoid over- and under diagnosis.

The double-blind, placebo-controlled, oral food challenge (DBPCFC) is considered the gold standard for diagnosing food allergy and it is preferred for research purposes [14]. The overall level of risk associated with food challenges has been examined. A retrospective series reviewed 584 OFCs performed in children who were estimated to have a ≤50% risk of reaction. Forty-three percent of the challenges were positive. Thirty-nine percent of the reactions were mild, 33% moderate, and 28% severe. The type and incidence of the different reactions were cutaneous (78%), gastrointestinal (43%), oral (26%), lower respiratory (26%), and upper respiratory (25%). No patients had cardiovascular symptoms [15].

Participants with positive and negative skin tests will proceed to oral challenge, as sensitization does not have a linear correlation with clinical allergy. Although the risk of a positive reaction to oral challenge with finned wine with chitosan is very low (severe seafood allergy is usually mediated by major shellfish allergen tropomyosin, not present in chitosan), for safety purposes the challenges will be performed in an appropriate setting, with CPR support available, medication and a doctor present at all times.

Potential Benefits It will allow for patients with shellfish allergy to be informed if they can safely ingest this wine. Furthermore, it will be needed as a public health measure as this information could be included in the wine labels.

STUDY OBJECTIVES

To investigate the safety of chitosan, as wine fining agent, in patients with severe allergy to shrimp.

Primary Outcome: Result of a DBPCFC with chitosan fined wine.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 and less than 65 years
* Willing to comply with all study procedures and available for the duration of the study;
* Diagnosed with shrimp allergy, based on clinical history, plus positive skin tests and/or positive IgE;
* Previous anaphylactic reaction to shrimp;
* Either sex and of any race
* Provide signed and dated informed consent form

Exclusion Criteria:

* Dermatological disease which precludes or alters the results of skin tests
* History of wine/alcohol intolerance
* Acquired or hereditary immunodeficiency
* Neoplasia
* Psychiatric disease
* FEV1<70%
* Taking any systemic medication that might interfere with the study and that is not possible to withdraw, namely oral corticosteroids or immunomodulators in the last 4 weeks, or antihistamines in the last 10 days
* Under beta-blockers or ACE inhibitors
* Presence of any significant illness that could interfere with the study or alter its results or increase the risk of anaphylaxis, such as systemic mastocytosis
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events to a Double Blind Placebo Controlled Food Challenge with chitosan fined wine | Participants will be followed until one to two hours after the end of the Food Challenge, an expected average of 6 to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luís P Amaral, MD, Principal Investigator — * Intern
Locations (2):
- Portugal (2):
  - Universidade de Aveiro, Aveiro
  - Serviço de Imunoalergologia Hospital São João, Porto

REFERENCES:
- [Derived] Amaral L, Silva D, Couto M, Nunes C, Rocha SM, Coimbra MA, Coimbra A, Moreira A. Safety of chitosan processed wine in shrimp allergic patients. Ann Allergy Asthma Immunol. 2016 May;116(5):462-3. doi: 10.1016/j.anai.2016.02.004. Epub 2016 Mar 19. No abstract available. PMID 27009439